CLINICAL TRIAL: NCT02158000
Title: Aspiration of Excessive Endometrial Fluid at the Day of Ovum Retrieval Plus Diosmin in (ICSI) Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid abd aziz mohamed, lecturer of ob/gyn, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: khalid-ahmed 5
Record Dates: First submitted 2014-06-05; First posted 2014-06-06 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Diosmin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): In group A , 100 women with excessive endometrial fluid by transvaginal ultrasound during ICSI cycles are allocated to receive one tab / 8 hs of Diosmin ( 500mg) beginning from the day of ovum retrieval and for 3 days (till the day of embro trasfer) in addition to aspiration of the fluid by an IUI catheter.
  Interventions: Other: group A
- Group B (No Intervention): In group B (control group) 100 women with excessive endometrial fluid by transvaginal ultrasound during ICSI cycles, no thing will be done

INTERVENTIONS:
Other: group A — one tab every 8 hs Diosmin ( 500mg) beginning from the day of ovum retrieval in addition to aspiration of the fluid by an IUI catheter
  Other Names: Daflon
  Arms: Group A

SUMMARY:
To notify the effect of aspiration of excessive endometrial fluid in addition to Diosmin in cases undergoing intracytoplasmic sperm injection (ICSI) cycles.

DETAILED DESCRIPTION:
Objectives: To notify the effect of aspiration of excessive endometrial fluid in addition to Diosmin in cases undergoing intracytoplasmic sperm injection (ICSI) cycles.

Study design: Prospective randomized controlled clinical trial.

Patients and Methods: 200 women with excessive endometrial fluid by transvaginal ultrasound during ICSI cycles are randomly scheduled into two equal groups. In group A, one tab every 8 hs Diosmin ( 500mg) beginning from the day of ovum retrieval in addition to aspiration of the fluid by an IUI catheter ; while in group B (control group), no thing is given or done. The main outcome measures are presence of the fluid on the day of embryo transfer and the pregnancy rate on those patients.

ELIGIBILITY:
Inclusion Criteria:

* women with excessive endometrial fluid by transvaginal ultrasound during ICSI cycles

Exclusion Criteria:

* none

Ages: 23 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
the pregnancy rate | is checked 16 days after embryos transfer
  is assessed by :serum hCG test Beta sub-unit of hCG (serum hCG test)

SECONDARY OUTCOMES:
presence of the fluid on the day of embryo transfer | at the day of embryo transfer
  detection of excessive endometrial fluid by transvaginal ultrasound during ICSI cycles

CONTACTS AND LOCATIONS:
Overall Officials: khalid mohamed, Study Chair — Department of Obstetrics and Gynecology, Benha University Hospital
Locations (1):
- Benha univesity hospital, Banhā, El Qualyobia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
on research gate

REFERENCES:
- [Derived] Saad AS, Mohamed KAA. Aspiration with Diosmin Intake in Endometrial Cavity Fluid Accumulation in ART Cycles: A Randomized Controlled Trial. J Obstet Gynaecol India. 2023 Aug;73(4):336-342. doi: 10.1007/s13224-023-01791-7. Epub 2023 Aug 31. PMID 37701088